CLINICAL TRIAL: NCT04493398
Title: Erythritol Air-polishing Versus Curette/Ultrasonic Debridement of Mandibular Furcation Lesions in Supportive Periodontal Therapy A 12-Month Randomized Controlled Trial
Brief Title: Air-polishing or Conventional Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Knut N. Leknes, Professor, University of Bergen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/793
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Periodontitis; Adult Periodontitis
Keywords: Furcation involvement; Periodontal maintenance
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized, single-masked controlled trial (RCT). A split-mouth study design where each of the furcation in the lower jaw molars was randomized to the two specific treatments. Hence, each patient received both interventions randomly allocated to each side of the lower jaw.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Two operators performed the clinical aspects of this study. Author TS, masked to treatment assignments, performed all clinical recordings and sampling, author IU performed all treatments. All analyses were performed by a statistician (SAL) who had not taken part in data collection or treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium curette and ultrasonic. (Active Comparator): Debridement of mandibular furcations with conventional ultrasonic/curette (control).
  Interventions: Procedure: Gracey curette.; Procedure: Ultrasonic scaler.
- Erythritol air-polishing. (Experimental): Treatment of mandibular furcations with erythritol powder/air-polishing system (test)
  Interventions: Procedure: Erythritol air-polishing.

INTERVENTIONS:
Procedure: Gracey curette. — Root planed was performed with curettes (Gracey SAS, Hu-Friedy, Chicago, IL, USA).
  Arms: Titanium curette and ultrasonic.
Procedure: Ultrasonic scaler. — Debridement was performed with an ultrasonic scaler (Piezon Master 400 Perio Slim Tip®; Electro Medical System, Nyon, Switzerland).
  Arms: Titanium curette and ultrasonic.
Procedure: Erythritol air-polishing. — Treatment was performed with a low abrasive erythritol powder (Air-flow powder plus®, EMS, Nyon, Switzerland ) applied through a Perio-Flow hand piece connected to an airflow unit (Air-Flow Master®, EMS, Nyon, Switzerland).
  Arms: Erythritol air-polishing.

SUMMARY:
Background: To effectively disrupt microbial biofilm and remove dental calculus with minimal damage to the root surface and soft tissues with limited patient discomfort constitute a significant tenet of periodontal therapy. The aim of the present prospective 12-month study was to compare clinical and microbiological effects following an erythritol air-polishing vs. conventional mechanical debridement of furcation defects in a cohort of periodontal maintenance patients.

Methods: Twenty patients with grade II mandibular molar furcation defects volunteered to enroll in this study. In a split-mouth design, two furcation sites in each patient were randomly assigned to either receive subgingival debridement using erythritol air-polishing (test) or conventional ultrasonic/curette debridement (control) at baseline, and at 3, 6, 9 and 12 months. Probing depth, clinical attachment level and bleeding on probing were recorded at 3-month intervals. Subgingival microbiological samples obtained at baseline, 6 and 12 months were analyzed using checkerboard DNA-DNA hybridization. Discomfort from treatment was scored at 12 months using a visual analogue scale.

DETAILED DESCRIPTION:
INTRODUCTION.Traditionally, periodontal debridement is accomplished using curettes, sonic or ultrasonic scalers, all presenting comparable outcomes.1,2 However, periodic root instrumentation may lead to dental hard tissue3-6 and soft tissue damage,7 and sensitivity due to exposure of dentinal tubules.8-10 Air-polishing using low abrasive glycine or trehalose powder has been shown to reach similar clinical outcomes as hand and ultrasonic instrumentation, but with less hard tissue loss.11-16 Moreover, air-polishing provides superior outcomes relative to patient comfort and time efficiency.7,11,12,14 Recently, a low abrasive erythritol powder with comparable physical properties to glycine air-polishing powder was introduced for subgingival air-polishing.17 Erythritol, a non-toxic, chemically neutral and completely water-soluble polyol is widely used in food industry as an artificial sweetener. Two studies comparing conventional mechanical debridement with erythritol air-polishing, reported similar results in supportive periodontal therapy (SPT) relative to clinical and microbiological outcomes.18,19 Such observations are also reflected in a systematic review concluding that air-polishing systems as a monotherapy are comparable to conventional therapy in patients undergoing SPT in single- and multi-rooted teeth without furcations.20 Moreover, inhibitory effects on pathogenic bacteria including Porphyromonas gingivalis have also been observed.21 To the investigator's knowledge, no prospective studies investigating the efficacy of a low abrasive erythritol air-polishing system in molar furcation defects during SPT have been reported. The objective of this 12-month prospective study was to compare clinical and microbiological effects following an erythritol air-polishing system vs. conventional mechanical debridement of furcation defects in a cohort of periodontal maintenance patients.

METHOD AND MATERIALS. The study protocol and informed consent following the Helsinki Declaration of 1975 (version 2008) was approved by the Medical Research Ethics Committee (2016/793), University of Bergen, Norway. Participating subjects read and signed the informed consent prior to enrolling in the study.

Prestudy calibration and training. Two operators performed the clinical aspects of this study. Author TS, masked to treatment assignments, performed all clinical recordings and sampling, author IU performed all treatments.

Sample size. The sample size estimation was based on change in PD. A difference of 0.5 mm was considered clinically relevant.22 Standard deviation of the difference between repeated PD measurements from the intra-calibration exercise was 0.5 mm. A power analysis based on 20 subjects and with the level of significance (α) set to 0.05, resulted in 98.9% power to detect a true difference of 0.5 mm.

Treatments. Following baseline examination, mandibular jaw quadrants were randomized (coin toss) to either receive debridement using the erythritol powder/air-polishing system (test) or conventional ultrasonic/curette instrumentation (control) using a split-mouth study design. Sequence of treatments was randomized in a similar fashion. Treatments were delivered at baseline, and repeated at 3, 6, 9 and 12 months. Test sites thus received root debridement using the low abrasive erythritol powder (Air-flow powder plus®, EMS, Nyon, Switzerland ) applied through a Perio-Flow hand piece connected to an airflow unit (Air-Flow Master®, EMS, Nyon, Switzerland). The hand piece was fitted with a nozzle for subgingival delivery directing the power/air jet perpendicular to the root surface at the water exit at the tip of the nozzle. The nozzle was inserted to the apical aspect of furcation sites with PD≥ 4 mm using striking movements over the furcation area for 5 sec.12 Sites adjoining the test site with PD≥ 4 mm were similarly treated.

Control sites were debrided using an ultrasonic scaler (Piezon Master 400 Perio Slim Tip®; Electro Medical System, Nyon, Switzerland) with power set at 75% and water as coolant, and root planed with sharp curettes (Gracey SAS, Hu-Friedy, Chicago, IL, USA).

Patients were returned to their regular SPT upon completion of study. Gingival crevicular fluid assessments. Gingival crevicular fluid (GCF) was recorded at baseline, and at 6 and 12 months. Briefly, furcation sites were isolated with cottons rolls, cleaned for supragingival plaque, and air-dried. A perio paper strip was then placed 1-2 mm into the orifice of the site and left in place for 30 sec. Next, the perio strip was inserted into the Periotron 8000® (Oraflow, Smithtown, NY, USA) calibrated to estimate the volume of GCF collected.

Microbiological assessments. At baseline, and at 6 and 12 months the supragingival area above the furcation site was wiped clean using sterile cotton pellets. Three sterile paper points were then inserted into the pocket of the furcation site. The paper points were kept in place 20 sec27 removed and immersed into pre-reduced, anaerobic transport medium (PRAS; Dental Transport Medium, Morgan Hill, CA, USA).

Pain experience assessments. Visual analogue scale (VAS) scores were used to estimate patient discomfort experienced during test and control treatment.31 Scoring was performed at 12 months following completion of the debridement with 0="no pain" and 100="worst pain I can imagine".

Statistical analysis Data were entered into MS-Excel (Microsoft, Redmond, WA, USA ) proofed for errors and then imported into Stata, version 15 (StataCorp, College Station, TX, USA).

Summary statistics (means ± SEM) for the clinical variables were calculated for the test and control at baseline, and at 6 and 12 months. Due to the repeated nature of data, a mixed effect model taking into consideration incomplete data at 12 months was applied to analyze the data at patient and tooth level. Time and treatment were considered fixed factors. Mixed models were applied for both primary and secondary outcome variables.

For testing differences in microbial composition at test and control sites harboring different proportions of bacteria >105 at baseline, and at 6 and 12 months, logistic regression models with robust standard error were applied. VAS scores were analyzed using ordinary linear regression models with robust standard error. The level of significance was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Received supportive periodontal therapy (SPT) every 3-6 months for 2-3 years following periodontal therapy.
2. Having bilateral non-mobile, fully erupted mandibular first, second or third molars with degree II furcation defects.
3. PD≥4 mm with bleeding or pus on probing. -

Exclusion Criteria:

1. Mobile mandibular molars, molars with clinical or radiographic evidence of supra-/subgingival calculus or apical pathology.
2. Use of systemic antibiotics within 6 months or SPT within 3 months of study.
3. Any current medical condition affecting periodontal treatment or use of the abrasive air-polishing device.
4. Subjects with diabetes, cancer, HIV/aids, acute infections, disorders that may compromise wound healing, or pregnant women.

   -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
In 20 patients with grade II mandibular molar furcation defects, probing depth (PD) will be measured. | 12 months.
  PD: The vertical distance from the gingival margin to the probable base of the pocket in mm.
In 20 patients with grade II mandibular molar furcation defects clinical attachment level (CAL) will be measured. | 12 months.
  CAL: The vertical distance in mm from the cemento-enamel junction or the margin of a dental restoration to the probable base of the pocket.

SECONDARY OUTCOMES:
Bleeding on probing (BoP). | 12 months.
  At site level, BoP was recorded as present upon gentle probing to the base of the vertical furcation pocket.
Gingival crevicular fluid (GCF). | 12 months.
  Twenty test and control sites were isolated with cottons rolls, cleaned for supragingival plaque, and air-dried. A perio paper strip was then placed 1-2 mm into the orifice of the site and left in place for 30 sec. The perio strip was inserted into the Periotron 8000® (Oraflow, Smithtown, NY, USA) calibrated to estimate the volume of GCF collected.
Visual analogue scale (VAS). | 12 months.
  VAS scores were used to estimate patient discomfort experienced during test and control treatment by drawing a vertical line on a 100-millimeter standardized horizontal line (0="no pain" and 100="worst pain I can imagine").

CONTACTS AND LOCATIONS:
Overall Officials: Knut N. Leknes, Professor, Principal Investigator — Department of Clinical Dentistry - Periodontics, University of Bergen, NORWAY.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson TG Jr. Supportive periodontal treatment introduction--definition, extent of need, therapeutic objectives, frequency and efficacy. Periodontol 2000. 1996 Oct;12:11-5. doi: 10.1111/j.1600-0757.1996.tb00074.x. No abstract available. PMID 9567987
- [Background] Badersten A, Nilveus R, Egelberg J. Effect of nonsurgical periodontal therapy. II. Severely advanced periodontitis. J Clin Periodontol. 1984 Jan;11(1):63-76. doi: 10.1111/j.1600-051x.1984.tb01309.x. PMID 6363463
- [Background] Zappa U, Smith B, Simona C, Graf H, Case D, Kim W. Root substance removal by scaling and root planing. J Periodontol. 1991 Dec;62(12):750-4. doi: 10.1902/jop.1991.62.12.750. PMID 1765938
- [Background] Flemmig TF, Petersilka GJ, Mehl A, Hickel R, Klaiber B. Working parameters of a magnetostrictive ultrasonic scaler influencing root substance removal in vitro. J Periodontol. 1998 May;69(5):547-53. doi: 10.1902/jop.1998.69.5.547. PMID 9623897
- [Background] Lie T, Leknes KN. Evaluation of the effect on root surfaces of air turbine scalers and ultrasonic instrumentation. J Periodontol. 1985 Sep;56(9):522-31. doi: 10.1902/jop.1985.56.9.522. PMID 3897504
- [Background] Schmidlin PR, Beuchat M, Busslinger A, Lehmann B, Lutz F. Tooth substance loss resulting from mechanical, sonic and ultrasonic root instrumentation assessed by liquid scintillation. J Clin Periodontol. 2001 Nov;28(11):1058-66. doi: 10.1034/j.1600-051x.2001.281111.x. PMID 11686828
- [Background] Petersilka GJ. Subgingival air-polishing in the treatment of periodontal biofilm infections. Periodontol 2000. 2011 Feb;55(1):124-42. doi: 10.1111/j.1600-0757.2010.00342.x. No abstract available. PMID 21134232
- [Background] Fischer C, Wennberg A, Fischer RG, Attstrom R. Clinical evaluation of pulp and dentine sensitivity after supragingival and subgingival scaling. Endod Dent Traumatol. 1991 Dec;7(6):259-65. doi: 10.1111/j.1600-9657.1991.tb00214.x. PMID 1820859
- [Background] Latheef P, Sirajuddin S, Gundapaneni V, Mn K, Apine A. Iatrogenic Damage to the Periodontium Caused by Periodontal Treatment Procedures. Open Dent J. 2015 Jun 26;9:203-7. doi: 10.2174/1874210601509010203. eCollection 2015. PMID 26312087
- [Background] Lin YH, Gillam DG. The Prevalence of Root Sensitivity following Periodontal Therapy: A Systematic Review. Int J Dent. 2012;2012:407023. doi: 10.1155/2012/407023. Epub 2012 Oct 31. PMID 23193405
- [Background] Petersilka GJ, Steinmann D, Haberlein I, Heinecke A, Flemmig TF. Subgingival plaque removal in buccal and lingual sites using a novel low abrasive air-polishing powder. J Clin Periodontol. 2003 Apr;30(4):328-33. doi: 10.1034/j.1600-051x.2003.00290.x. PMID 12694431
- [Background] Petersilka G. Re: "Subgingival plaque removal using a new air-polishing device". Moene R, Decaillet F, Andersen E, Mombelli A. (J Periodontol 2010;81:79-88.). J Periodontol. 2010 Jul;81(7):962-3. doi: 10.1902/jop.2010.100118. No abstract available. PMID 20553116
- [Background] Flemmig TF, Arushanov D, Daubert D, Rothen M, Mueller G, Leroux BG. Randomized controlled trial assessing efficacy and safety of glycine powder air polishing in moderate-to-deep periodontal pockets. J Periodontol. 2012 Apr;83(4):444-52. doi: 10.1902/jop.2011.110367. Epub 2011 Aug 23. PMID 21861637
- [Background] Wennstrom JL, Dahlen G, Ramberg P. Subgingival debridement of periodontal pockets by air polishing in comparison with ultrasonic instrumentation during maintenance therapy. J Clin Periodontol. 2011 Sep;38(9):820-7. doi: 10.1111/j.1600-051X.2011.01751.x. Epub 2011 Jul 7. PMID 21736599
- [Background] Caygur A, Albaba MR, Berberoglu A, Yilmaz HG. Efficacy of glycine powder air-polishing combined with scaling and root planing in the treatment of periodontitis and halitosis: A randomised clinical study. J Int Med Res. 2017 Jun;45(3):1168-1174. doi: 10.1177/0300060517705540. Epub 2017 Apr 20. PMID 28425827
- [Background] Kruse AB, Akakpo DL, Maamar R, Woelber JP, Al-Ahmad A, Vach K, Ratka-Krueger P. Trehalose powder for subgingival air-polishing during periodontal maintenance therapy: A randomized controlled trial. J Periodontol. 2019 Mar;90(3):263-270. doi: 10.1002/JPER.17-0403. Epub 2018 Nov 9. PMID 30311948
- [Background] Hagi TT, Hofmanner P, Salvi GE, Ramseier CA, Sculean A. Clinical outcomes following subgingival application of a novel erythritol powder by means of air polishing in supportive periodontal therapy: a randomized, controlled clinical study. Quintessence Int. 2013 Nov-Dec;44(10):753-61. doi: 10.3290/j.qi.a30606. PMID 24078975
- [Background] Hagi TT, Hofmanner P, Eick S, Donnet M, Salvi GE, Sculean A, Ramseier CA. The effects of erythritol air-polishing powder on microbiologic and clinical outcomes during supportive periodontal therapy: Six-month results of a randomized controlled clinical trial. Quintessence Int. 2015 Jan;46(1):31-41. doi: 10.3290/j.qi.a32817. PMID 25262675
- [Background] Muller N, Moene R, Cancela JA, Mombelli A. Subgingival air-polishing with erythritol during periodontal maintenance: randomized clinical trial of twelve months. J Clin Periodontol. 2014 Sep;41(9):883-9. doi: 10.1111/jcpe.12289. Epub 2014 Aug 7. PMID 25041441
- [Background] Ng E, Byun R, Spahr A, Divnic-Resnik T. The efficacy of air polishing devices in supportive periodontal therapy: A systematic review and meta-analysis. Quintessence Int. 2018;49(6):453-467. doi: 10.3290/j.qi.a40341. PMID 29700503
- [Background] Hashino E, Kuboniwa M, Alghamdi SA, Yamaguchi M, Yamamoto R, Cho H, Amano A. Erythritol alters microstructure and metabolomic profiles of biofilm composed of Streptococcus gordonii and Porphyromonas gingivalis. Mol Oral Microbiol. 2013 Dec;28(6):435-51. doi: 10.1111/omi.12037. Epub 2013 Jul 29. PMID 23890177
- [Background] Bunaes DF, Lie SA, Enersen M, Aastrom AN, Mustafa K, Leknes KN. Site-specific treatment outcome in smokers following non-surgical and surgical periodontal therapy. J Clin Periodontol. 2015 Oct;42(10):933-42. doi: 10.1111/jcpe.12462. Epub 2015 Oct 28. PMID 26407817
- [Background] Muhlemann HR, Son S. Gingival sulcus bleeding--a leading symptom in initial gingivitis. Helv Odontol Acta. 1971 Oct;15(2):107-13. No abstract available. PMID 5315729
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Hamp SE, Nyman S, Lindhe J. Periodontal treatment of multirooted teeth. Results after 5 years. J Clin Periodontol. 1975 Aug;2(3):126-35. doi: 10.1111/j.1600-051x.1975.tb01734.x. PMID 1058213
- [Background] Barros SP, Williams R, Offenbacher S, Morelli T. Gingival crevicular fluid as a source of biomarkers for periodontitis. Periodontol 2000. 2016 Feb;70(1):53-64. doi: 10.1111/prd.12107. PMID 26662482
- [Background] Belibasakis GN, Schmidlin PR, Sahrmann P. Molecular microbiological evaluation of subgingival biofilm sampling by paper point and curette. APMIS. 2014 Apr;122(4):347-52. doi: 10.1111/apm.12151. Epub 2013 Jul 24. PMID 23879704
- [Background] Socransky SS, Haffajee AD, Smith C, Martin L, Haffajee JA, Uzel NG, Goodson JM. Use of checkerboard DNA-DNA hybridization to study complex microbial ecosystems. Oral Microbiol Immunol. 2004 Dec;19(6):352-62. doi: 10.1111/j.1399-302x.2004.00168.x. PMID 15491460
- [Background] Socransky SS, Smith C, Martin L, Paster BJ, Dewhirst FE, Levin AE. "Checkerboard" DNA-DNA hybridization. Biotechniques. 1994 Oct;17(4):788-92. PMID 7833043
- [Background] Socransky SS, Haffajee AD, Cugini MA, Smith C, Kent RL Jr. Microbial complexes in subgingival plaque. J Clin Periodontol. 1998 Feb;25(2):134-44. doi: 10.1111/j.1600-051x.1998.tb02419.x. PMID 9495612
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Krohn-Dale I, Boe OE, Enersen M, Leknes KN. Er:YAG laser in the treatment of periodontal sites with recurring chronic inflammation: a 12-month randomized, controlled clinical trial. J Clin Periodontol. 2012 Aug;39(8):745-52. doi: 10.1111/j.1600-051X.2012.01912.x. Epub 2012 Jun 13. PMID 22694321
- [Background] Hujoel PP, Loesche WJ. Efficiency of split-mouth designs. J Clin Periodontol. 1990 Nov;17(10):722-8. doi: 10.1111/j.1600-051x.1990.tb01060.x. PMID 2262586
- [Background] Hujoel PP, DeRouen TA. Validity issues in split-mouth trials. J Clin Periodontol. 1992 Oct;19(9 Pt 1):625-7. doi: 10.1111/j.1600-051x.1992.tb01709.x. PMID 1430289
- [Background] Hujoel PP. Design and analysis issues in split mouth clinical trials. Community Dent Oral Epidemiol. 1998 Apr;26(2):85-6. doi: 10.1111/j.1600-0528.1998.tb01932.x. No abstract available. PMID 9645400
- [Background] Cobb CM. Non-surgical pocket therapy: mechanical. Ann Periodontol. 1996 Nov;1(1):443-90. doi: 10.1902/annals.1996.1.1.443. No abstract available. PMID 9118268
- [Background] Bower RC. Furcation morphology relative to periodontal treatment. Furcation entrance architecture. J Periodontol. 1979 Jan;50(1):23-7. doi: 10.1902/jop.1979.50.1.23. PMID 283222
- [Background] Bower RC. Furcation morphology relative to periodontal treatment. Furcation root surface anatomy. J Periodontol. 1979 Jul;50(7):366-74. doi: 10.1902/jop.1979.50.7.366. No abstract available. PMID 288913
- [Background] Petersilka GJ, Tunkel J, Barakos K, Heinecke A, Haberlein I, Flemmig TF. Subgingival plaque removal at interdental sites using a low-abrasive air polishing powder. J Periodontol. 2003 Mar;74(3):307-11. doi: 10.1902/jop.2003.74.3.307. PMID 12710749
- [Background] Armitage GC. Analysis of gingival crevice fluid and risk of progression of periodontitis. Periodontol 2000. 2004;34:109-19. doi: 10.1046/j.0906-6713.2002.003427.x. No abstract available. PMID 14717858
- [Background] Tsang YC, Corbet EF, Jin LJ. Subgingival glycine powder air-polishing as an additional approach to nonsurgical periodontal therapy in subjects with untreated chronic periodontitis. J Periodontal Res. 2018 Jun;53(3):440-445. doi: 10.1111/jre.12532. Epub 2018 Mar 25. PMID 29574763
- [Background] Bunaes DF, Mustafa M, Mohamed HG, Lie SA, Leknes KN. The effect of smoking on inflammatory and bone remodeling markers in gingival crevicular fluid and subgingival microbiota following periodontal therapy. J Periodontal Res. 2017 Aug;52(4):713-724. doi: 10.1111/jre.12438. Epub 2017 Mar 17. PMID 28306142
- [Background] Hagi TT, Klemensberger S, Bereiter R, Nietzsche S, Cosgarea R, Flury S, Lussi A, Sculean A, Eick S. A Biofilm Pocket Model to Evaluate Different Non-Surgical Periodontal Treatment Modalities in Terms of Biofilm Removal and Reformation, Surface Alterations and Attachment of Periodontal Ligament Fibroblasts. PLoS One. 2015 Jun 29;10(6):e0131056. doi: 10.1371/journal.pone.0131056. eCollection 2015. PMID 26121365
- [Background] Antczak-Bouckoms AA, Tulloch JF, Berkey CS. Split-mouth and cross-over designs in dental research. J Clin Periodontol. 1990 Aug;17(7 Pt 1):446-53. doi: 10.1111/j.1600-051x.1990.tb02343.x. PMID 2201705
- [Derived] Ulvik IM, Saethre T, Bunaes DF, Lie SA, Enersen M, Leknes KN. A 12-month randomized controlled trial evaluating erythritol air-polishing versus curette/ultrasonic debridement of mandibular furcations in supportive periodontal therapy. BMC Oral Health. 2021 Jan 21;21(1):38. doi: 10.1186/s12903-021-01397-3. PMID 33478480